CLINICAL TRIAL: NCT00614055
Title: A 16 Week Randomised, Open Labelled, 3 Armed, Parallel Group, Treat-to-target Trial Comparing Once Daily Injection of SIAC 30 (B), SIAC 45 (B) and Insulin Glargine, All in Combination With Metformin in Subjects With Type 2 Diabetes Failing on OAD Treatment
Brief Title: Comparison of Two NN5401 Formulations Versus Insulin Glargine, All in Combination With Metformin in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN5401-1791; 2007-002476-33 (EudraCT Number)
Record Dates: First submitted 2008-01-30; First posted 2008-02-13 (Estimated); Results first posted 2015-11-17 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin degludec, insulin aspart drug combination; Insulin Glargine; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Insulin glargine (Active Comparator)
  Interventions: Drug: insulin glargine; Drug: metformin
- SIAC 30 (B) (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart; Drug: metformin
- SIAC 45 (B) (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart; Drug: metformin

INTERVENTIONS:
Drug: insulin degludec/insulin aspart — Formulation 1: Treat-to-target dose titration scheme, injection s.c., once daily
  Arms: SIAC 30 (B)
Drug: insulin degludec/insulin aspart — Formulation 2: Treat-to-target dose titration scheme, injection s.c., once daily
  Arms: SIAC 45 (B)
Drug: insulin glargine — Treat-to-target dose titration scheme, injection s.c., once daily
  Arms: Insulin glargine
Drug: metformin — Tablets, 1500-2000 mg/day

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to compare two NN5401 (SIAC, insulin degludec/insulin aspart) formulations with each other and with insulin glargine, all in combination with metformin in insulin naive subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. (Trial-related activities are any procedure that would not have been performed during normal management of the subject.)
* Insulin naïve type 2 diabetes subjects (as diagnosed clinically) for at least 3 months (no previous insulin treatment or previous short term insulin treatment maximum 14 days within the last 3 months)
* Treatment with one or two oral anti-diabetic drugs (OADs): metformin, sulfonylurea, other insulin secretagogue (e.g. repaglinide, nateglinide), alpha-glucosidase inhibitors for at least 2 month at a stable maximum tolerated dose or at least half maximum allowed dose according to locally approved summary of product characteristics (SPC)
* HbA1c, 7.0 - 11.0 % (both inclusive)
* Body Mass Index (BMI), 25.0 - 37.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* Metformin contraindication according to local practice
* Thiazolidinedione (TZD) treatments within the previous three months prior to Visit 1
* Any systemic treatment with products, which in the investigator's opinion could interfere with glucose or lipid metabolism (e.g. systemic corticosteroids) within 3 months prior to randomisation
* Subject has a clinically significant, active (during the past 12 months) disease of the gastrointestinal, pulmonary, neurological, genitourinary, or haematological system that, in the opinion of the investigator, may confound the results of the trial or pose additional risk in administering trial product

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2008-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (24):
- France (6):
  - Novo Nordisk Investigational Site, Alès
  - Novo Nordisk Investigational Site, Brest
  - Novo Nordisk Investigational Site, La Rochelle
  - Novo Nordisk Investigational Site, Le Creusot
  - Novo Nordisk Investigational Site, Mont-de-Marsan
  - Novo Nordisk Investigational Site, Vénissieux
- Germany (6):
  - Novo Nordisk Investigational Site, Bad Kreuznach
  - Novo Nordisk Investigational Site, Bad Mergentheim
  - Novo Nordisk Investigational Site, Dormagen
  - Novo Nordisk Investigational Site, Hohenmölsen
  - Novo Nordisk Investigational Site, Neuss
  - Novo Nordisk Investigational Site, Neuwied
- Norway (6):
  - Novo Nordisk Investigational Site, Elverum
  - Novo Nordisk Investigational Site, Hamar
  - Novo Nordisk Investigational Site, Kongsvinger
  - Novo Nordisk Investigational Site, Oslo
  - Novo Nordisk Investigational Site, Stavanger
  - Novo Nordisk Investigational Site, Tromsø
- Novo Nordisk Investigational Site, Bucharest, Romania
- Spain (5):
  - Novo Nordisk Investigational Site, Almería
  - Novo Nordisk Investigational Site, Partida de Bacarot
  - Novo Nordisk Investigational Site, Seville
  - Novo Nordisk Investigational Site, Valencia
  - Novo Nordisk Investigational Site, Valladolid

REFERENCES:
- [Result] Heise T, Tack CJ, Cuddihy R, Davidson J, Gouet D, Liebl A, Romero E, Mersebach H, Dykiel P, Jorde R. A new-generation ultra-long-acting basal insulin with a bolus boost compared with insulin glargine in insulin-naive people with type 2 diabetes: a randomized, controlled trial. Diabetes Care. 2011 Mar;34(3):669-74. doi: 10.2337/dc10-1905. Epub 2011 Feb 1. PMID 21285389
- [Result] Ma Z, Parkner T, Christiansen JS, Laursen T. IDegAsp: a novel soluble insulin analogs combination. Expert Opin Biol Ther. 2012 Nov;12(11):1533-40. doi: 10.1517/14712598.2012.722203. Epub 2012 Sep 4. PMID 22946603
- [Result] Liebl A, Davidson J, Mersebach H, Dykiel P, Tack CJ, Heise T. A novel insulin combination of insulin degludec and insulin aspart achieves a more stable overnight glucose profile than insulin glargine: results from continuous glucose monitoring in a proof-of-concept trial. J Diabetes Sci Technol. 2013 Sep 1;7(5):1328-36. doi: 10.1177/193229681300700524. PMID 24124961
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 22 sites in 5 countries: France (4 sites), Germany (5 sites), Norway (5 sites), Romania (3 sites) and Spain (5 sites).
Pre-assignment Details: During a run-in period of 2 weeks, metformin was up-titrated to 1500/ 2000 mg/day, which was maintained for 1 week. Subjects who tolerated the metformin dose for a week and had a median of 3 self measured glucose values before breakfast, on 3 consecutive days before randomisation, of ≥ 7.5 mmol/l, were randomised to 1 of the 3 treatment groups
Groups:
- SIAC 30 (B): Soluble insulin analogue combination 30 (SIAC 30, 70 volume percent insulin degludec, 600 nmol/ml and 30 volume percent insulin aspart, 600 nmol/ml; formulation B) was given subcutaneously once daily (OD) before dinner in combination with at least 1500 mg/day metformin (tablets) for 16 weeks. Insulin doses were individually adjusted.
- SIAC 45 (B): Soluble insulin analogue combination 45 (SIAC 45, 55 volume percent insulin degludec, 600 nmol/ml and 45 volume percent insulin aspart, 600 nmol/ml; formulation B) was given subcutaneously once daily (OD) before dinner in combination with at least 1500 mg/day metformin (tablets) for 16 weeks. Insulin doses were individually adjusted.
- Insulin Glargine: Insulin glargine was given subcutaneously once daily (OD) before dinner in combination with at least 1500 mg/day metformin (tablets) for 16 weeks. Insulin doses were individually adjusted.
Period: Overall Study
Arm/Group | SIAC 30 (B) | SIAC 45 (B) | Insulin Glargine
Started | 59 | 59 | 60
Exposed | 59 | 59 | 60
Completed | 55 | 53 | 55
Not Completed | 4 | 6 | 5
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Protocol Violation | 2 | 2 | 1
Not completed — Lack of Efficacy | 0 | 0 | 2
Not completed — Unclassified | 1 | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SIAC 30 (B) | SIAC 45 (B) | Insulin Glargine | Total
Number analyzed (Participants) | 59 | 59 | 60 | 178
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (8.8) | 60.2 (8.4) | 58.4 (8.4) | 59.1 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 25 | 16 | 63
  Male | 37 | 34 | 44 | 115
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.3 (1.2) | 8.6 (1.5) | 8.4 (1.3) | 8.5 (1.3)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 11.1 (3.3) | 11.5 (3.2) | 12.1 (3.5) | 11.6 (3.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Haemoglobin (HbA1c)
Description: Change from baseline in HbA1c after 16 weeks of treatment
Time Frame: Week 0, Week 16
Population: Full analysis set (FAS) included all randomised subjects and missing data was imputed using last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | SIAC 30 (B) | SIAC 45 (B) | Insulin Glargine
Number analyzed (Participants) | 59 | 59 | 60
percentage of glycosylated haemoglobin | -1.31 (1.01) | -1.46 (1.39) | -1.29 (1.10)

2. Secondary Outcome: Change in Fasting Plasma Glucose (FPG)
Description: Change from baseline in FPG after 16 weeks of treatment
Time Frame: Week 0, Week 16
Population: The FAS included all randomised subjects and missing data was imputed using LOCF.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | SIAC 30 (B) | SIAC 45 (B) | Insulin Glargine
Number analyzed (Participants) | 59 | 59 | 60
mmol/L | -4.30 (3.45) | -4.10 (3.09) | -5.07 (3.85)

3. Secondary Outcome: Mean of 9-point Self Measured Plasma Glucose Profile (SMPG)
Description: Mean of SMPG after 16 weeks of treatment. Plasma glucose measured: before breakfast, 120 minutes after start of breakfast, before lunch, 120 minutes after start of lunch, before dinner, 120 minutes after start of dinner, bedtime, at 4 am and before breakfast.
Time Frame: Week 16
Population: The FAS included all randomised subjects and missing data was imputed using LOCF.
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | SIAC 30 (B) | SIAC 45 (B) | Insulin Glargine
Number analyzed (Participants) | 59 | 59 | 60
mmol/L | 8.34 (0.75) | 8.31 (0.78) | 8.42 (0.78)

4. Secondary Outcome: Rate of Treatment Emergent Adverse Events (AEs)
Description: Corresponds to rate of AEs per 100 patient years of exposure. Severity assessed by investigator. Mild: no or transient symptoms, no interference with subject's daily activities. Moderate: marked symptoms, moderate interference with subject's daily activities. Severe: considerable interference with subject's daily activities, unacceptable. Serious AE: AE that at any dose results in any of the following: death, a life-threatening experience, in-subject hospitalization/prolongation of existing hospitalisation, persistent/significant disability/incapacity/congenital anomaly/birth defect.
Time Frame: Week 0 to Week 16 + 5 days follow up
Population: Safety analysis set (SAS) included all subjects who received at least one dose of the investigational product or its comparator.
Measure: Number; unit: Events/100 years of patient exposure
Arm/Group | SIAC 30 (B) | SIAC 45 (B) | Insulin Glargine
Number analyzed (Participants) | 59 | 59 | 60
Events/100 years of patient exposure
  Adverse events (AEs) | 441 | 310 | 295
  Serious AEs | 11 | 6 | 0
  Severe AEs | 6 | 0 | 0
  Moderate AEs | 138 | 123 | 61
  Mild AEs | 298 | 187 | 234
  Fatal AEs | 0 | 0 | 0

5. Secondary Outcome: Rate of Major and Minor Hypoglycaemic Episodes
Description: Rate of Major and Minor hypoglycaemic episodes per 100 patient years of exposure (PYE). Major if unable to treat her/himself. Minor if able to treat her/himself and plasma glucose below 3.1 mmol/L.
Time Frame: Week 0 to Week 16 + 5 days follow up
Population: The FAS included all randomised subjects.
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | SIAC 30 (B) | SIAC 45 (B) | Insulin Glargine
Number analyzed (Participants) | 59 | 59 | 60
Episodes/100 years of patient exposure
  Major | 0 | 0 | 0
  Minor | 115 | 240 | 67

6. Secondary Outcome: Rate of Nocturnal Major and Minor Hypoglycaemic Episodes
Description: Rate of nocturnal Major and Minor hypoglycaemic episodes per 100 patient years of exposure (PYE). Major if unable to treat her/himself. Minor if able to treat her/himself and plasma glucose below 3.1 mmol/L. Episodes were defined as nocturnal if the time of onset was between 23:00 (included) and 06:00 (excluded).
Time Frame: Week 0 to Week 16 + 5 days follow up
Population: The FAS included all randomised subjects.
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | SIAC 30 (B) | SIAC 45 (B) | Insulin Glargine
Number analyzed (Participants) | 59 | 59 | 60
Episodes/100 years of patient exposure
  Major | 0 | 0 | 0
  Minor | 6 | 158 | 17

7. Secondary Outcome: Laboratory Safety Parameters (Biochemistry): Alanine Aminotransferase (ALAT)
Description: Values at screening (Week -4) and at Week 16
Time Frame: Week -4, Week 16
Population: The SAS included all subjects who received at least one dose of the investigational product or its comparator.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | SIAC 30 (B) | SIAC 45 (B) | Insulin Glargine
Number analyzed (Participants) | 59 | 59 | 60
IU/L
  Week -4 , N=58, 59, 60 | 31.9 (18.3) | 29.7 (15.3) | 33.7 (23.1)
  Week 16 , N=54, 54, 57 | 23.9 (13.1) | 23.2 (9.7) | 22.3 (10.3)

8. Secondary Outcome: Laboratory Safety Parameters (Biochemistry): Aspartate Aminotransferase (ASAT)
Description: Values at screening (Week -4) and at Week 16
Time Frame: Week -4, Week 16
Population: The SAS included all subjects who received at least one dose of the investigational product or its comparator.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | SIAC 30 (B) | SIAC 45 (B) | Insulin Glargine
Number analyzed (Participants) | 59 | 59 | 60
IU/L
  Week -4, N=58, 59, 60 | 24.8 (14.6) | 22.0 (8.3) | 24.0 (14.1)
  Week 16, N=54, 54, 57 | 21.1 (8.2) | 20.0 (5.8) | 19.2 (6.4)

9. Secondary Outcome: Laboratory Safety Parameters (Biochemistry): Serum Creatinine
Description: Values at screening (Week -4) and at Week 16
Time Frame: Week -4, Week 16
Population: The SAS included all subjects who received at least one dose of the investigational product or its comparator.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | SIAC 30 (B) | SIAC 45 (B) | Insulin Glargine
Number analyzed (Participants) | 59 | 59 | 60
umol/L
  Week -4 , N=58, 59, 60 | 76.4 (15.4) | 75.8 (14.4) | 77.4 (13.9)
  Week 16 , N=54, 54, 57 | 75.7 (15.4) | 74.9 (15.6) | 76.8 (14.6)

10. Secondary Outcome: Vital Signs: Diastolic Blood Pressure (BP)
Description: Values at baseline (Week 0) and at Week 16
Time Frame: Week 0, Week 16
Population: The SAS included all subjects who received at least one dose of the investigational product or its comparator.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SIAC 30 (B) | SIAC 45 (B) | Insulin Glargine
Number analyzed (Participants) | 59 | 59 | 60
mmHg
  Week 0 (Baseline), N=59, 59, 60 | 78 (8) | 78 (8) | 79 (8)
  Week 16, N=56, 53, 58 | 76 (8) | 77 (9) | 77 (7)

11. Secondary Outcome: Vital Signs: Systolic Blood Pressure (BP)
Description: Values at baseline (Week 0) and at Week 16
Time Frame: Week 0, Week 16
Population: The SAS included all subjects who received at least one dose of the investigational product or its comparator.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SIAC 30 (B) | SIAC 45 (B) | Insulin Glargine
Number analyzed (Participants) | 59 | 59 | 60
mmHg
  Week 0 (Baseline), N=59, 59, 60 | 135 (15) | 133 (14) | 135 (15)
  Week 16, N=56, 53, 58 | 129 (13) | 133 (12) | 129 (12)

12. Secondary Outcome: Vital Signs: Pulse
Description: Values at baseline (Week 0) and at Week 16
Time Frame: Week 0, Week 16
Population: The SAS included all subjects who received at least one dose of the investigational product or its comparator.
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | SIAC 30 (B) | SIAC 45 (B) | Insulin Glargine
Number analyzed (Participants) | 59 | 59 | 60
beats/minute
  Week 0 (Baseline), N=59, 59, 60 | 73 (10) | 75 (10) | 75 (9)
  Week 16, N=56, 53, 58 | 71 (10) | 69 (9) | 71 (11)

13. Secondary Outcome: Physical Examination
Description: Physical examination is performed at baseline (Week 0) and after 8 and 16 weeks of treatment. If any new findings or deterioration in previous findings were observed during the trial, these were recorded as AEs and are therefore not presented separately as no analysis was performed.
Time Frame: Week 0, Week 8, Week 16
Arm/Group | Insulin Glargine | SIAC 30 (B) | SIAC 45 (B)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: The adverse events were collected in a time frame of 16 weeks + 7 days follow up
Description: The SAS included all subjects who received at least one dose of the investigational product or its comparator.
Arm/Group | SIAC 30 (B) | SIAC 45 (B) | Insulin Glargine
Serious Adverse Events (participants affected / at risk) | 2/59 | 1/59 | 0/60
Other Adverse Events (participants affected / at risk) | 23/59 | 16/59 | 13/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SIAC 30 (B) (N=59) | SIAC 45 (B) (N=59) | Insulin Glargine (N=60)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SIAC 30 (B) (N=59) | SIAC 45 (B) (N=59) | Insulin Glargine (N=60)
Dyspepsia (Gastrointestinal disorders) | 3 (4) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 3 (3)
Nasopharyngitis (Infections and infestations) | 4 (4) | 3 (3) | 1 (3)
C-reactive protein increased (Investigations) | 14 (14) | 5 (5) | 9 (9)
Dyslipidaemia (Metabolism and nutrition disorders) | 6 (6) | 4 (4) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.